CLINICAL TRIAL: NCT06204926
Title: Diagnostic Efficacy of Convolutional Neural Network Based Algorithm in Predicting Intraoperative Complications and Postoperative Outcomes in Small Incision Lenticule Extraction
Brief Title: Diagnostic Efficacy of CNN in Predicting Intraoperative Complications and Postoperative Outcomes in SMILE
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Collaborators: Hangzhou Huaxia Eye Hospital (Unknown); Nanchang Bright Eye Hospital (Unknown)
Responsible Party: Principal Investigator, Jian Xiong, Associate research fellow; Attending physician, Second Affiliated Hospital of Nanchang University
Other Study IDs: [2023] No.(96)
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-01

CONDITIONS: Deep Convolutional Neural Network; Small-incision Lenticule Extraction (SMILE) Surgery; Intraoperative Complications; Postoperative Outcomes
Keywords: femtosecond laser small-incision lenticule extraction; Intraoperative Complications; Deep Convolutional Neural Network; Postoperative Outcomes
MeSH Terms: conditions — Smiling; Intraoperative Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Eyes with SMILE surgeries: Eyes with SMILE surgeries which were performed by surgeons with experiences.
  Interventions: Diagnostic Test: AI diagnostic algorithm

INTERVENTIONS:
Diagnostic Test: AI diagnostic algorithm — The SMILE procedures collected would be assessed by the algorithm. The performance of the algorithm would be assessed, including accuracy, AUC, sensitivity and specificity.

SUMMARY:
To evaluate the diagnostic efficiency of the neural network in predicting complications of Small Incision Lenticule Extraction in a multi-center cross-sectional study.

DETAILED DESCRIPTION:
The primary cause of global visual impairment currently is refractive error, and Small Incision Lenticule Extraction (SMILE) using femtosecond laser for corneal stromal lenticule extraction can alter the refractive power. However, complications such as opaque bubble layer (OBL), negative pressure detachment, and black spots may arise during the SMILE laser scanning process due to individual differences in corneal characteristics, significantly affecting the normal course of surgery and postoperative recovery. Experienced docters can often predict intraoperative complications based on scan images, patient cooperation, and other factors, but the learning curve is relatively long. At present, artificial intelligence has achieved the accuracy comparable to human physicians in the interpretation of medical imaging of many different diseases.Previously, we have trained a deep convolutional neural network for predicting intraoperative complications in SMILE procedures. The current multi-center study is designed to evaluate the efficacy of the convolutional neural network based algorithm in predicting intraoperative complications and to assess its utility in the real world.

ELIGIBILITY:
Inclusion Criteria:

* A condition in which the spherical equivalent refractive error of an eye is ≤-0.50 D when ocular accommodation is relaxed;
* Age ≥18 years;
* Spherical equivalent (SE) ≥-10.0D;
* Corrected distance visual acuity (CDVA) ≥16/20;
* Stable myopia for at least 2 years;
* No contact lenses wearing for at least 2 weeks.

Exclusion Criteria:

* The presence or history of eye conditions other than myopia and astigmatism, such as keratoconus or external eye injury;
* A history of eye surgery;
* The presence or history of systemic diseases.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients from clinics in different eye centers across China. Each subject must with complete surgical video recording and medical records.
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
AUROC of convolutional neural network in predicting OBL area | Day 0
  The area under the receiver operating characteristic of convolutional neural network in predicting opaque bubble layer area during the SMILE surgeries
AUROC of convolutional neural network in predicting progressive suction loss | Day 0
  The area under the receiver operating characteristic of convolutional neural network in predicting progressive suction loss during the SMILE surgeries
AUROC of convolutional neural network in predicting effective optical zone | Day 7
  The area under the receiver operating characteristic of convolutional neural network in predicting effective optical zone after the SMILE surgeries

SECONDARY OUTCOMES:
Sensitivity and specificity of convolutional neural network in predicting OBL area | Day 0
  Sensitivity and specificity of convolutional neural network in predicting opaque bubble layer area during the SMILE surgeries
Sensitivity and specificity of convolutional neural network in predicting progressive suction loss | Day 0
  Sensitivity and specificity of convolutional neural network in predicting progressive suction loss during the SMILE surgeries
Sensitivity and specificity of convolutional neural network in predicting effective optical zone | Day 7, Day 30, Day 90
  ensitivity and specificity of convolutional neural network in predicting effective optical zone after the SMILE surgeries

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No